CLINICAL TRIAL: NCT07035457
Title: Relative Bioavailability of Single Doses of Vicadrostat and Empagliflozin Administered Alone Compared to Combined Administration to Healthy Male Subjects (an Open Label, Randomised, Three-way Crossover Trial)
Brief Title: A Study in Healthy Men to Compare the Amount of Vicadrostat and Empagliflozin in the Blood When Taken Separately and Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1378-0024; 2024-518103-21-00 (Registry Identifier: CTIS); U1111-1313-3279 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment sequence A: R1-R2-T (Experimental): Reference 1 (R1): vicadrostat Reference 2 (R2): empagliflozin Test (T): vicadrostat and empagliflozin taken together
  Interventions: Drug: Vicadrostat; Drug: Jardiance®
- Treatment sequence B: R2-T-R1 (Experimental): Reference 1 (R1): vicadrostat Reference 2 (R2): empagliflozin Test (T): vicadrostat and empagliflozin taken together
  Interventions: Drug: Vicadrostat; Drug: Jardiance®
- Treatment sequence C: T-R1-R2 (Experimental): Reference 1 (R1): vicadrostat Reference 2 (R2): empagliflozin Test (T): vicadrostat and empagliflozin taken together
  Interventions: Drug: Vicadrostat; Drug: Jardiance®

INTERVENTIONS:
Drug: Vicadrostat — Vicadrostat
  Other Names: BI 690517
Drug: Jardiance® — Jardiance®
  Other Names: Empagliflozin

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of vicadrostat and empagliflozin when administered in combination or individually.

ELIGIBILITY:
Inclusion Criteria :

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with international council for harmonisation-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria :

* Any finding in the medical examination (including ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 105 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 65 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of vicadrostat in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Reference 1 (Days 1, 2 and 3), Test (Days 1, 2 and 3)
Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Reference 2 (Days 1, 2, 3 and 4), Test (Days 1, 2, 3 and 4)
Maximum measured concentration of vicadrostat in plasma (Cmax) | Reference 1 (Days 1, 2 and 3), Test (Days 1, 2 and 3)
Maximum measured concentration of empagliflozin in plasma (Cmax) | Reference 2 (Days 1, 2, 3 and 4), Test (Days 1, 2, 3 and 4)

SECONDARY OUTCOMES:
Area under the concentration-time curve of vicadrostat in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz ) | Reference 1 (Days 1, 2 and 3), Test (Days 1, 2 and 3)
Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Reference 2 (Days 1, 2, 3 and 4), Test (Days 1, 2, 3 and 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com